CLINICAL TRIAL: NCT02503644
Title: A Randomized, Double-blind, Placebo-controlled, Multicentre Proof-of-concept Trial of IVA337 in the Treatment of Diffuse Cutaneous Systemic Sclerosis
Brief Title: Proof-of-concept Trial of IVA337 in Diffuse Cutaneous Systemic Sclerosis
Acronym: FASST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVA_01_337_HSSC_15_001
Record Dates: First submitted 2015-06-30; First posted 2015-07-21 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Scleroderma, Diffuse; Diffuse Cutaneous Systemic Sclerosis
Keywords: diffuse cutaneous systemic sclerosis; scleroderma; IVA337; dcSSc; lanifibranor
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — lanifibranor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IVA337 800mg (Active Comparator): Patients receive twice daily 400mg IVA337.
  Interventions: Drug: IVA337
- IVA337 1200mg (Active Comparator): Patients receive twice daily 600mg IVA337.
  Interventions: Drug: IVA337
- Placebo (Placebo Comparator): Patients receive twice daily placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IVA337 — Capsules of 200mg IVA337
  Other Names: lanifibranor
  Arms: IVA337 1200mg; IVA337 800mg
Drug: Placebo — Identical capsules without active substance
  Other Names: No other names at present
  Arms: Placebo

SUMMARY:
Systemic sclerosis (SSc), or scleroderma is a connective tissue disease of autoimmune origin. It is a life-threatening orphan disease with severe physical and psychosocial consequences. IVA337 has a novel mechanism of action and this study is designed to compare IVA337 at two dose levels with a placebo control treatment. Patients will be unaware of the treatment they are receiving and will be randomized to one of three treatment arms , either IVA337 400mg bid, IVA337 600mg bid or placebo bid. They will receive drug for 48 weeks and during that time assessments will be made to monitor both the efficacy and safety of the treatment.

DETAILED DESCRIPTION:
Study design: randomized, double-blind, placebo-controlled, multicentre phase 2 proof-of-concept trial of IVA337 for the treatment DcSSc.

The treatments are randomly assigned. The randomisation is stratified for background therapy to ensure even distribution of background therapies among treatment groups.

There are 3 parallel treatment groups: placebo, IVA337 400mg bid and IVA337 600mg bid (identical capsules of 200mg IVA337 or placebo). Both, patient and investigator are blinded.

The treatment lasts 48 weeks. A follow-up assessment takes place 4 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent documented by signature
* Systemic sclerosis according to ACR/EULAR 2103 criteria (van de Hoogen 2013)
* Diffuse cutaneous SSc subset according to LeRoy's criteria
* Diagnosis within the past 3 years as defined by the first non-Raynaud's symptom
* MRSS between 10 and 25
* Age between 18 and 75, male or female

Patients on stable treatment (for >3 months) with prednisone ≤ 10 mg, methotrexate≤ 20 mg/w, azathioprine ≤ 150 mg/d, mycophenolate mofetil ≤ 2g/d, or leflunomide ≤ 20 mg/d may be included in the study; the therapy must be maintained as background therapy.

Exclusion Criteria:

* Cyclophosphamide during the past 3 months
* Requirement of IV prostanoids for pulmonary hypertension in the last 3 months
* Renal insufficiency defined by a creatinine clearance of less than 30 ml/min (CKD-EPI or MDRD formula) and/or past/current renal crisis
* Hepatic impairment i.e. primary biliary cirrhosis and unexplained persistent liver function abnormality,
* Gallbladder disease (Cholelithiasis is not an exclusion criterion)
* Diabetic ketoacidosis
* Severe cardiac (LVEF <45%) and/or pulmonary disease (FVC < 50% or pulmonary hypertension proven by right heart catheterisation)
* History of heart failure, symptomatic coronary artery disease, significant ventricular tachyarrhythmia, stent placement, coronary artery bypass surgery, and/or myocardial infarction.
* Recipient of solid organ transplant
* Gastrointestinal involvement preventing oral administration of study drug
* Chronic infections, positive serology for infection with hepatitis B or C.
* Pregnancy, Lactation. Woman of childbearing potential unwilling to use a medically acceptable form of birth control
* History of malignancy within the last 5 years, except for resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ cervical cancer
* A recent history of alcohol or drug abuse, non-compliance with other medical therapies
* Participation in a clinical study involving another investigational drug or device within 4 weeks before the Pre-treatment Visit
* Laboratory parameters at the pre-treatment visit showing any of the following abnormal results: transaminases > 2x the upper limit of normal (ULN) and/or bilirubin > 2x ULN; neutrophil count < 1,500/mm3; platelet count < 100,000/mm3; haemoglobin < 9 g/dL
* Known hypersensitivity or allergy to class of drugs or the investigational product
* Any condition or treatment, which in the opinion of the investigator, places the subject at unacceptable risk as a patient in the trial
* Co-therapy with biologics: Wash-out period: Any anti-TNF agent in the last 3-months: adalimumab, certolizumab, etanercept, golimumab, infliximab; abatacept and tocilizumab in the last 3 months; rituximab in the last 6 months.
* Any other significant heart disease or any clinically significant ECG abnormality reported by central ECG reading.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Measurement of skin thickness by the Modified Rodnan Skin Score (MRSS) | 48 weeks
  Mean change of the MRSS from baseline

SECONDARY OUTCOMES:
Response rates based on MRSS improvement | 12, 24, 32, 48 weeks
  MRSS response rates:
  Initial definition: improvers are defined by a reduction ≥5 points and ≥25 % of MRSS; Additional definition: improvers are defined by a reduction
  ≥ 4 points and ≥ 20% of MRSS based on Quillinan et al. (2014, 2017)
Overall progression of the disease: defined as absence of rescue therapy and absence of severe organ involvement | 28, 32,40, and 48 weeks
  Overall progression of the disease: defined as absence of rescue therapy and absence of severe organ involvement
Lung function measured by FVC% predicted | 24 and 48 weeks
  Change in pulmonary function
Lung function by cDLCO% predicted | 24 and 48 weeks
  Change in pulmonary function
Scleroderma Health Assessment Questionnaire (SHAQ) | 24 and 48 weeks
  Changes in patient reported outcomes
Gastrointestinal tract symptoms severity and its impact on patients' well-being assessed by the UCLA SCTC GIT | 24 and 48 weeks
  Changes in patient reported outcomes
Patient-reported health status assessed by PROMIS29 | 24 and 48 weeks
  Changes in patient reported outcomes
Physical and mental health assessed by SF36 | 24 and 48 weeks
  Changes in patient reported outcomes
Digital ulcer net burden (defined as total number of ulcers at a certain time point minus number of ulcers at baseline) and proportion of patients who do not develop new ulcers | 12, 24, 32 and 48 weeks
  Digital ulcer net burden (defined as total number of ulcers at a certain time point minus number of ulcers at baseline) and proportion of patients who do not develop new ulcers
Hand function assessed by the Cochin Hand Function Scale | 12, 24, 32 and 48 weeks
  Hand function assessed by the Cochin Hand Function Scale
Patient global assessment of disease activity assessed by a visual analogue scale | 24 and 48 weeks
  Patient global assessments of disease activity (VAS)
Physician global assessment of disease activity assessed by a visual analogue scale | 24 and 48 weeks
  Physician global assessment of disease activity (VAS)
Change in the Combined Response Index for Systemic Sclerosis (CRISS) | 24 and 48 weeks
  Composed of five variables: MRSS, FVC % predicted, physician and patient global assessments, and HAQ-DI score
Percent of patients who need escape therapy | 28, 32,40, and 48 weeks
  Need for escape therapy
Percent of patients who experience a new severe organ involvement | 2, 4, 8,12, 16, 24, 28, 32, 40, 48, and 52 weeks
  Severe organ involvement
Number of participants with adverse events as a measure of safety and tolerability | 2, 4, 8, 12, 16, 20, 24, 28, 32, 40, 44, 48, and 52 weeks
  Frequency and type of AEs
Routine and specific laboratory tests (composite) to assess safety and tolerability | 2, 12, 20, 24, 32, 36, 44, 48, and 52 weeks
  creatine kinase, N-terminal pro-brain natriuretic peptide, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, γ-glutamyl transferase, total bilirubin, direct bilirubin,RBC and WBC count, reticulocytes, haemoglobin, haematocrit, albumin , Quick, aPTT, INR, BUN, plasma creatinine, microalbuminuria, homocysteine, urinalysis (dip stick), glycated haemoglobin, creatine phosphokinase increase, platelet counts, plasma osteocalcin, serum beta C-terminal telopeptide (β-CTx or B-Crosslaps), Differential: neutrophils, eosinophils, basophils, monocytes, lymphocytes, cholesterol, triglycerides, albumin, total protein, C-reactive protein (CRP), adiponectin, serology HIV and hepatitis infection: Hep. A antibodies, B antibodies and antigen, C antibodies, serum b-HCG.

OTHER OUTCOMES:
Raynaud attacks assessed by a diary and the Raynaud condition score (VAS) | Daily during week 9 and week 25
Progression of the disease assessed by changes of the activity of specific SSc biomarkers in the blood | 12, 24, and 48 weeks
  Mean changes in activity biomarkers
Progression of the disease assessed by changes of the activity of specific SSc biomarkers in the skin | 48 weeks
  Mean changes in activity biomarkers
Population pharmacokinetics to confirm the pharmacokinetic profile, including Cmax, Tmax, AUC, half-life (t1/2), clearance (CL/F) and volume of distribution (Vd/F) | 2, 24, and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Allanore, Professor, Principal Investigator — Université Paris Descartes, Hôpital Cochin, Service de Rhumatologie A & INSERM, Paris, France,; Christopher Denton, Professor, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (49):
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski, Pleven
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - University Multiprofile Hospital for Active Treatment -Kaspela, Plovdiv
  - University Multiprofile Hospital for Active Treatment - "Sveti Ivan Rilski", Sofia
- France (4):
  - Hôpital Pellegrin, Bordeaux
  - CHRU de Lille- Hôpital Claude Huriez, Lille
  - Hopital Cochin, Paris
  - University Hospital of Strasbourg, Strasbourg
- Germany (10):
  - Kerckhoff-Klinik, Bad Nauheim
  - Charité- Universitätsmedizin Berlin, Berlin
  - Chaité-Universtätsmedezin Berlin, Berlin
  - Klinik fur Dermatologie und Venerologie der Universitat zu Köln, Cologne
  - Univertaetsklinikum Carl Gustav Carus, Dresden
  - University of Erlangen-Nuremberg, Erlangen
  - CIRI GmbH Centrum für Innovative Diagnostik und Therapie, Frankfurt
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Kilinik für Hautkrankenheiten, Münster
  - Universtätsklinik Ulm, Ulm
- Italy (9):
  - Istituto di Clinica Medica Generale Polo Didattico, Ancona
  - Azienda Ospedalaria Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Salvatore ASL L'Aquila, L’Aquila
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - University of Padova, Padua
  - Ospedale di Alta Specializzazione "San Camillo", Roma
  - Policlinico Umberto I, Roma
  - Universita degli Studi de Verona, Verona
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus MC Universitair Medisch Centrum Rotterdam, Rotterdam
- Poland (6):
  - Centrum Miriada Prywatny, Bialystok
  - University Hospital in Bydgoszcz, Bydgoszcz
  - CM Plejady, Krakow
  - Reumed, Lublin
  - Medycine Centrum Hetmanska Poznan, Poznan
  - Centrum Medyczne Oporow, Wroclaw
- Slovenia (2):
  - University Medical centre Ljubljana, Ljubljana
  - University Medical Centre Maribor, Maribor
- Spain (8):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hopital Universitario Gregorio Marañon, Madrid
  - Hopital 12 de Octubre, Madrid
  - Hopital Universitario Sanchinarro, Madrid
  - Hospital La Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Dr Peset, Valencia
- Switzerland (2):
  - University Hospital Lausanne, Lausanne
  - University Hospital Zurich, Zurich
- United Kingdom (2):
  - Leeds Institut of Rheumatic and Musculoskeletal Medicine, Leeds
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No